CLINICAL TRIAL: NCT04991194
Title: Effect of Age-gender on the Pharmacokinetic and Pharmacodynamic Profiles of BIA 5 1058. An Open-label, Parallel Group, Multiple Dose 10-day Study.
Brief Title: Effect of Age-gender on the Pharmacokinetic and Pharmacodynamic Profiles of BIA 5 1058
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-51058-105; 2015-003682-28 (EudraCT Number)
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — zamicastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIA 5-1058 1200 mg (Part I) (Experimental): Subjects received 1200 mg of BIA 5-1058 once a day (od), in fasting conditions, for 10 days
  Interventions: Drug: BIA 5-1058
- BIA 5-1058 400 mg (Part II) (Experimental): Subjects received 400 mg of BIA 5-1058 od, in fasting conditions, for 10 days.
  Interventions: Drug: BIA 5-1058

INTERVENTIONS:
Drug: BIA 5-1058 — Each subject was administered either 1200 mg (Part 1) or 400 mg (Part 2) BIA 5-1058 od for 10 days, in fasting conditions for 8 hours [Day (D)2 to D9] or 10 hours (D1 and D13), and remained fasted for 2 hours (D2 to D9) or 4 hours (D1 and D13) post-dose. The formulation was tablets 100 mg and the mode of administration was oral.
  Other Names: Zamicastat

SUMMARY:
the purpose of this study is to determine the effect of age on the Pharmacokinetics (PK) profile of BIA 5-1058 at steady state after multiple oral doses

DETAILED DESCRIPTION:
This was a single-centre, open-label, parallel group, non-randomised, two-part multiple dose 10-day study in healthy young and elderly male and female subjects. The study comprised a screening evaluation between 2 and 28 days before the first Investigational Medicinal Product (IMP) administration, a hospitalisation period of 15 days comprising a treatment period of 10 days, and a follow-up visit approximately 7 days after discharge.

Part 1: Subjects received 1200 mg of BIA 5-1058 once a day (od), in fasting conditions, for 10 days Part 2 : Subjects received 400 mg of BIA 5-1058 od, in fasting conditions, for 10 days.

ELIGIBILITY:
Inclusion Criteria:

All subjects (young and elderly):

1. A signed and dated informed consent form before any study-specific screening procedure was performed;
2. Healthy male and female subjects as determined by the Investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs and digital 12-lead electrocardiogram (ECG);
3. Non-smoker or ex-smokers for at least 3 months at screening;
4. BMI between 18 and 30 kg/m2, inclusive;
5. Negative tests for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus antibodies (HCV Ab) and anti-human immunodeficiency virus antibodies (HIV-1 and HIV-2 Ab) at screening;
6. Clinical laboratory test results clinically acceptable at screening and admission to the study;
7. Negative screen for alcohol and drugs of abuse at screening and admission to the study;

   If male:
8. Using an effective method of contraception with a pregnant partner or partner of childbearing potential (condom or occlusive cap [diaphragm or cervical or vault caps] with spermicidal foam or gel or film or cream or suppository; true abstinence; or vasectomy) throughout the study;
9. Refraining from donating sperm throughout the study.

   Young subjects only:
10. Males and females aged between 18 and 40 years, inclusive.

    If female:
11. No childbearing potential by reason of surgery or at least 1 year post-menopause (i.e., 12 months post last menstrual period), or menopause confirmed by follicle-stimulating hormone (FSH) testing;
12. If of childbearing potential, using an effective non-hormonal method of contraception [intrauterine device or intrauterine system; condom or occlusive cap (diaphragm or cervical or vault caps) with spermicidal foam or gel or film or cream or suppository; true abstinence; or vasectomized male partner, provided that he is the sole partner of that subject] for all the duration of the study;
13. If of childbearing potential, negative serum pregnancy test at screening and negative urine pregnancy test on admission to the study.

    Elderly subjects only:
14. Males and females older than 65 years, inclusive.

Exclusion Criteria:

All subjects (young and elderly):

1. Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders;
2. Clinically relevant surgical history;
3. History of relevant atopy or drug hypersensitivity;
4. History of alcoholism or drug abuse;
5. Consumption of more than 14 units of alcohol a week [1 unit corresponds to 1 glass of 12° wine (10 cL), 1 glass of 45° pastis (2.5 cL), 1 glass of 40° whisky (2.5 cL), 1 glass of 12° champagne (10 cL), 1 glass of 18°aperitif drink (7 cL) or one 25-cL glass of 5°beer];
6. Significant infection or known inflammatory process at screening or admission to study;
7. Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to the study;
8. Previous use of BIA 5-1058;
9. Use of any investigational drug or participation in any clinical trial within 90 days prior to screening;
10. Participation in more than 2 clinical trials within the 12 months prior to screening;
11. Donation or reception of any blood or blood products within the 3 months prior to screening;
12. Vegetarians, vegans or other medical dietary restrictions;
13. Not able to communicate reliably with the Investigator;
14. Unlikely to co-operate with the requirements of the study.

    If male:
15. Not using an accepted effective method of contraception;
16. Refusing to refrain from donating sperm throughout the study.

    Young subjects only:
17. Use of medicines within 2 weeks of admission that could affect the safety or other study assessments, in the Investigator's opinion;

    If female of childbearing potential:
18. Pregnant or breastfeeding;
19. Not using an accepted effective contraceptive method or using oral contraceptives.

    Elderly subjects only:
20. For elderly subjects, previously prescribed medications that interfered with absorption, distribution, metabolism, and excretion or safety/tolerability evaluation of BIA 5-1058 and adrenal or renal function were prohibited; however, previously prescribed medications that did not interfere with absorption, distribution, metabolism, and excretion or safety/tolerability evaluation of BIA 5-1058, adrenal or renal function and which could not interfere with the objectives of the study were allowed if the dose regimen had been stable for at least 4 weeks and was expected to remain stable throughout the study. Such concomitant medications were to be reviewed and mutually agreed upon by the Sponsor and the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 4 weeks
  Pharmacokinetic analysis
  Blood samples for PK analysis were taken at the following times:
  On D1: before BIA 5-1058 dosing (pre-dose), and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 h post-dose (before the second administration on D2).
  On D3, D7, D8 and D9: before BIA 5-1058 dosing. From D10 to D13: before BIA 5-1058 dosing, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 (D11), 36 (D11), 48 (D12), 60 (D12) and 72h post-dose (D13).
Time of occurrence of Cmax (tmax) | Up to 4 weeks
  Pharmacokinetic analysis
  Blood samples for PK analysis were taken at the following times:
  On D1: before BIA 5-1058 dosing (pre-dose), and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 h post-dose (before the second administration on D2).
  On D3, D7, D8 and D9: before BIA 5-1058 dosing. From D10 to D13: before BIA 5-1058 dosing, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 (D11), 36 (D11), 48 (D12), 60 (D12) and 72h post-dose (D13).
Area under the plasma concentration-time curve (AUC) from time zero to the last sampling time at which the drug concentration was at or above the lower limit of quantification (AUC0-t) | Up to 4 weeks
  Pharmacokinetic analysis
  Blood samples for PK analysis were taken at the following times:
  On D1: before BIA 5-1058 dosing (pre-dose), and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 h post-dose (before the second administration on D2).
  On D3, D7, D8 and D9: before BIA 5-1058 dosing. From D10 to D13: before BIA 5-1058 dosing, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 (D11), 36 (D11), 48 (D12), 60 (D12) and 72h post-dose (D13).
Area under the plasma concentration-time curve from time zero to 24 hours after last dosing (AUC0-24) | Up to 4 weeks
  Pharmacokinetic analysis
  Blood samples for PK analysis were taken at the following times:
  On D1: before BIA 5-1058 dosing (pre-dose), and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 h post-dose (before the second administration on D2).
  On D3, D7, D8 and D9: before BIA 5-1058 dosing. From D10 to D13: before BIA 5-1058 dosing, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 (D11), 36 (D11), 48 (D12), 60 (D12) and 72h post-dose (D13).
Apparent terminal half-life (t½) | Up to 4 weeks
  Pharmacokinetic analysis
  Blood samples for PK analysis were taken at the following times:
  On D1: before BIA 5-1058 dosing (pre-dose), and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 h post-dose (before the second administration on D2).
  On D3, D7, D8 and D9: before BIA 5-1058 dosing. From D10 to D13: before BIA 5-1058 dosing, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 (D11), 36 (D11), 48 (D12), 60 (D12) and 72h post-dose (D13).
Apparent total body clearance (CL/F) | Up to 4 weeks
  Pharmacokinetic analysis
  Blood samples for PK analysis were taken at the following times:
  On D1: before BIA 5-1058 dosing (pre-dose), and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 h post-dose (before the second administration on D2).
  On D3, D7, D8 and D9: before BIA 5-1058 dosing. From D10 to D13: before BIA 5-1058 dosing, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 (D11), 36 (D11), 48 (D12), 60 (D12) and 72h post-dose (D13).

IPD SHARING:
Plan to Share IPD: Undecided